CLINICAL TRIAL: NCT07364032
Title: A Randomized Controlled Trial Comparing a Mindfulness-based Program With Standard Therapeutic Follow-up During Pregnancy: Effects on Maternal Well-being, Infant Outcomes, and Mother-Infant Attachment
Brief Title: Comparison Between a Mindfulness-Based Program and Standard Therapeutic Follow-Up During Pregnancy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universite Cote d'Azur (Other)
Responsible Party: Principal Investigator, Clara Beauvois, PhD Student, Universite Cote d'Azur
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CB-PCG-2022; ANR-15-IDEX-01 (Other Grant/Funding Number: Agence Nationale de la Recherche)
Record Dates: First submitted 2025-12-09; First posted 2026-01-23 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Mindfulness Protocols; Pregnancy
MeSH Terms: interventions — Referral and Consultation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness program (Experimental)
  Interventions: Behavioral: Mindfulness program
- Classical (Sham Comparator)
  Interventions: Other: Consultations

INTERVENTIONS:
Behavioral: Mindfulness program — 6 weeks of mindfulness
  Arms: Mindfulness program
Other: Consultations — 6 week of consultation with 1 consultation per week
  Arms: Classical

SUMMARY:
This study aims to evaluate the effects of a 6-week mindfulness meditation program in pregnant women, compared with a psychological support control program.

Participants in the mindfulness arm will complete one instructor-led meditation session per week and five guided audio meditation sessions at home each week.

The primary objectives are to determine whether the mindfulness program leads to:

Reduced negative affect, including stress, anxiety, depression, and sleep disturbances during pregnancy.

Increased positive affect, such as mindfulness skills, self-efficacy, happiness, and life satisfaction.

Enhanced maternal-fetal attachment during pregnancy and improved maternal-infant attachment one month postpartum.

Improved mother-infant interaction quality at 3 months postpartum.

More secure infant attachment at 12 months.

Better infant outcomes, including reduced crying intensity/duration at 1 and 3 months, and improved sleep quality at 12 months.

Overall, the study evaluates whether the mindfulness program provides greater benefits than a standard parenting support intervention.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women between 3 and 7.5 months of gestation (12-28 weeks).
* Ability to speak and read French sufficient to understand study documents and complete questionnaires.
* Willingness to participate in the study and to be randomized to one of the study groups.

Exclusion Criteria:

* Loss of the baby
* Participation in other prenatal support programs, including prenatal yoga, haptonomy, sophrology, or mindfulness courses.
* Severe or unstable psychiatric disorder. Inability to understand French or complete study questionnaires.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 70 (Estimated)
Dates: Start 2023-03-31 (Actual); Primary Completion 2026-08-30 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
Anxiety | Questionnaire will be completed at day 0 and 6 weeks later.
  French version of Pregnancy Related Anxiety Questionnaire (Reymond et al., 2020)
Stress | Questionnaire will be completed at day 0 and 6 weeks later.
  French version of Short Stress scale (Cungi et al., 2003)
Depression | Questionnaire will be completed at day 0 and 6 weeks later.
  French version of Edinburgh Postnatal Depression Scale, (Cox et al., 1987)
Sleep disorders | Questionnaire will be completed at day 0 and 6 weeks later.
  French version of The Pittsburgh sleep quality index, (Buysse et al., 1989)
Mindfulness | Questionnaire will be completed at day 0 and 6 weeks later.
  French version of Mindfulness Scale (Brown et Ryan., 2003)
Self efficacy | Questionnaire will be completed at day 0 and 6 weeks later.
  French version of Generalized Self-Efficacy scale (Schwarzer et al., 1995)
Happiness | Questionnaire will be completed at day 0 and 6 weeks later.
  French version of Subjective Happiness Scale (Lyubomirsky & Lepper, 1997)
Satisfaction of life | Questionnaire will be completed at day 0 and 6 weeks later.
  French version of The Satisfaction with Life Scale (Diener et al., 1985)
Prenatal Attachment | Questionnaire will be completed at day 0 and 6 weeks later.
  French version of Prenatal Attachment Inventory, (Muller, 1993)

SECONDARY OUTCOMES:
Cries of the baby | Questionnaires will be completed daily up to 1 and 3 months post partum
  French Version Colic infant questionnaire (Bellaiche et al., 2021)
Sleep disturbances | Questionnaires will be completed at 1 year Post partum
  French Version Sleep disturbance scale for children, (Lecuelle et al., 2020)
Post natal attachment | video at 1 year
  French version of Baby Interaction Scale (Beaupuy. 2021) Pediatric Infant Parent Exam (PIPE, Fiese et al., 2001)

CONTACTS AND LOCATIONS:
Locations (1):
- Clara Beauvois Cabinet de psychologie, Mouans-Sartoux, France

IPD SHARING:
Plan to Share IPD: Undecided